CLINICAL TRIAL: NCT03278652
Title: Use of Analgesic Drugs in Renal Colic in Emergency Room
Acronym: NEPHROPAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3033_NEPHROPAIN
Record Dates: First submitted 2017-09-05; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Renal Colic
MeSH Terms: conditions — Renal Colic | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with renal colic
  Interventions: Other: Consumption of drugs for analgesic use

INTERVENTIONS:
Other: Consumption of drugs for analgesic use — * Regular assessment of pain
  * Drug data will be collected (name, dosage, route of administration, time of delivery)

SUMMARY:
A prospective non-interventional study on the use of analgesic drugs in renal colic in emergency rooms

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Suspicion of renal colic (pain in a lumbar pit radiating to the external genital organs, rapidly progressive onset, non-febrile)

Exclusion Criteria:

* Shock
* Glasgow score less than 15
* Oxygen saturation less than 93% in ambient air
* Signs of intracranial hypertension (headache associated with vomiting)
* Suspicion of pneumothorax
* History of emphysema or chronic obstructive pulmonary disease
* Diving accident or suspicion of gas embolism
* Trauma of the face of interest in the area of application of the mask
* Abdominal gas distension
* Contraindication in Nonsteroidal anti-inflammatory drugs
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with renal colic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-04-19 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of analgesic drug used in the context of renal colic in emergency rooms by following the recommended and validated service protocol | During hospitalisation in emergency rooms
  Collection of name, dosage, route of administration, time of issue of the drug

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No